CLINICAL TRIAL: NCT01855880
Title: Efficacy, Safety, Tolerability, and Pharmacokinetics of Multiple Doses of AbGn-168H Administered by Intravenous Infusion to Patients With Moderate to Severe Chronic Plaque Psoriasis (Randomised, Double-blind, Placebo-controlled)
Brief Title: Phase IIa Study of Multiple Doses of AbGn-168H by iv Infusion in Moderate to Severe Chronic Plaque Psoriasis Patients
Acronym: AbGn-168H
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbGenomics B.V Taiwan Branch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012.005.01
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-04

CONDITIONS: Moderate to Severe Chronic Plaque Psoriasis
Keywords: psoriasis; dermatology; monoclonal antibody
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AbGn-168H Low Dose (Experimental): Subject to receive low dose of AbGn-168H intravenously
  Interventions: Biological: AbGn-168H
- AbGn-168H: High Dose (Experimental): Subject to receive high dose of AbGn-168H intravenously
  Interventions: Biological: AbGn-168H
- Placebo AbGn-168H (Placebo Comparator): Subject to receive placebo
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: AbGn-168H
  Arms: AbGn-168H Low Dose; AbGn-168H: High Dose
Biological: placebo
  Arms: Placebo AbGn-168H

SUMMARY:
This is a Phase IIa, randomised, double-blind, placebo-controlled, multiple dose, multi-center study of AbGn-168H in subjects with moderate to severe chronic plaque psoriasis.The objectives of this study is to investigate efficacy, safety, tolerability, and pharmacokinetics (PK) of multiple doses of AbGn-168H administered intravenously to patients with moderate to severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 (inclusive), males or females
2. Body weight < 140 kg
3. Patients with stable moderate to severe plaque-type psoriasis, no significant changes within the past 6 months, involving ≥ 10% body surface area, with disease severity PASI ≥ 10 at screening visit and visit 2, with at least 1 lesion for target lesion assessment.
4. Psoriasis disease duration of at least 6 months prior to screening
5. Patients must be candidates for systemic psoriasis treatment or phototherapy
6. Patient must give informed consent and sign an approved consent form prior to any study procedures
7. Females of childbearing potential must have a negative pregnancy test result prior to enrollment and agree to use a highly effective method of birth control during the study. A highly effective method of birth control is defined as one which results in a low failure rate (less than 1% per year).

Exclusion Criteria:

1. Patients with primary guttatae, erythrodermic, or pustular psoriasis and patients with drug-induced psoriasis
2. Evidence of current or previous clinically significant disease, medical condition other than psoriasis, or finding of the medical examination (including vital signs and ECG), that in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data. This criterion provides an opportunity for the investigator to exclude patients based on clinical judgment, even if other eligibility criteria are satisfied. (Psoriatic arthritis is not considered an exclusion)
3. HIV infection or a known HIV-related Malignancy.
4. Chronic or acute hepatitis B and C, or carrier status. Patient with anti-HBc Ab and undetectable anti-HBs Ab should also be excluded.
5. Tuberculosis, or a positive Tuberculin Skin Test (TST) for tuberculosis. Subjects previously received BCG vaccination can participate in the study after showing negative responses in Interferon-Gamma Release Assays (IGRA).
6. History of malignancy in the past 5 years or suspicion of active malignant disease except treated cutaneous squamous cell or basal cell carcinoma and carcinoma in situ of the cervix uteri.
7. History of allergy/hypersensitivity to a systemically administered biologic agent or its excipients
8. Use of biologic agents or investigational drug within 12 weeks prior to treatment, systemic anti-psoriatic medications or phototherapy within 4 weeks prior to treatment, or topical anti-psoriasis medications (except emollients) within 2 weeks prior to treatment
9. Intake of restricted medications (c.f. Section 4.2.2) or other drugs considered likely to interfere with the safe conduct of the study
10. History of alcohol abuse
11. History of drug abuse or positive drug screen at screening visit. Subjects with legitimate medically supervised uses of the drugs which are not excluded for other reasons (section 4.2.2 of the protocol) can be enrolled.
12. Any blood donation or significant blood loss within 4 weeks prior to Visit 2
13. Excessive (e.g. competitive) physical activities (within 1 week prior to administration or during the trial)
14. Patients with any of the following laboratory values at screening and are considered clinically significant by the investigators:

    * Haemoglobin, hematocrit, white blood cell count, absolute lymphocyte or neutrophil count, or platelet count < LLN (below the lower limit of the reference normal range)
    * ALT, AST and/or total bilirubin > 2.5xULN
    * Serum creatinine > 1.5x ULN

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
PASI75 | the achievement of at least 75% reduction from baseline PASI score (PASI75) at week 12 in each patient.
  The primary objective of this study is to investigate efficacy (clinical proof of concept) of AbGn-168H in patients with moderate to severe chronic plaque psoriasis following intravenous administration of multiple doses compared to placebo. In this trial, the high dose and low dose of AbGn-168 and placebo is administered weekly.

SECONDARY OUTCOMES:
safety and tolerability | At different time point for 16 weeks after the first treatment
  Safety measurements including physical examination, vital signs, ECG, clinical laboratory tests and adverse events
pharmacokinetics | At different time point for16 weeks after the first treatment
  AUC, Cmax, tmax, t1/2, MRT and Vss; additional parameters as needed

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Yao Lin, MD, PhD, Study Director — AbGenomics B.V Taiwan Branch; Mark Lebwohl, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (15):
- United States (15):
  - Baptist Health Certer for Clinical Research, Little Rock, Arkansas
  - Northwest AR Clinical Trials, Rogers, Arkansas
  - Visions Clinical Research, Boynton Beach, Florida
  - Renstar Medical Research, Ocala, Florida
  - Progressive Medical Research, Orange, Florida
  - Olympian Clinical Research, Tampa, Florida
  - DawesFretzin Clinical Research Group, LLC., Indianaopoli, Indiana
  - Indiana University Dermatology, Indianapolis, Indiana
  - Comprehensive Clinical Research, Berlin, New Jersey
  - University Urology Associates & Manhattan Research Associates, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Research Affiliation, Oklahoma City, Oklahoma
  - Radiant Research, Inc., Greer, South Carolina
  - Suzanne Bruce and Associates, The Center for Skin Research, Huston, Texas
  - West End Dermatology Assotiate, Richmond, Virginia